CLINICAL TRIAL: NCT00002450
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study of the Safety and Efficacy of Tenofovir Disoproxil Fumarate in Combination With Other Antiretroviral Agents for the Treatment of HIV-1 Infected Patients
Brief Title: Safety and Effectiveness of Tenofovir Disoproxil Fumarate (Tenofovir DF) Plus Other Anti-HIV Drugs in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 283D; GS-99-907
Record Dates: First submitted 2000-01-17; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-07

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Drug Administration Schedule; RNA, Viral; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate

SUMMARY:
The purpose of this study is to see if giving tenofovir DF plus a combination of other anti-HIV drugs is safe and effective.

DETAILED DESCRIPTION:
Patients are randomized 2:1 to add tenofovir DF once daily or placebo to their existing antiretroviral regimen in a blinded manner. Patients are stratified according to HIV-1 RNA level, CD4 cell count, and number of antiretroviral drugs taken prior to study entry. Patients and physicians are strongly discouraged from making changes in their antiviral therapies for at least 24 weeks post-randomization. After Week 24, changes in background antiretroviral therapy are permitted. At 24 weeks post-randomization, patients randomized to receive placebo are crossed over to receive open-label tenofovir DF once daily for the remainder of the 48-week study. While on study drug, patients are monitored for safety using periodic physical examinations and serial laboratory tests. Additionally, changes in plasma HIV RNA levels and CD4 cell counts are monitored to assess antiviral efficacy. At the end of the 48-week study period, patients are rolled over into extended dosing until tenofovir DF is commercially available or Gilead Sciences terminates the study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have been on stable anti-HIV therapy for at least 8 weeks with no more than 4 anti-HIV drugs at the time of study entry.
* Have a viral load (level of HIV in the blood) between 400 and 10,000 copies/ml.
* Have good kidney function.
* Are 18 to 65 years old.
* Agree to use a barrier method of birth control (such as condoms) during the study and for 30 days after.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a new AIDS-related illness diagnosed within 30 days of study entry.
* Have any other serious medical conditions, including kidney or bone disease, an active infection requiring antibiotics, or cancer (other than Kaposi's sarcoma or certain skin cancers).
* Have received a vaccine within 30 days of study entry.
* Are unable to take medications by mouth.
* Have ever taken tenofovir or adefovir dipivoxil.
* Have taken certain medications within 30 days of study entry, such as chemotherapy, corticosteroids, medications that affect the kidneys, treatment for Kaposi's sarcoma, or certain experimental drugs.
* Abuse alcohol or drugs.
* Are pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600

CONTACTS AND LOCATIONS:
Locations (61):
- United States (58):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Body Positive, Phoenix, Arizona
  - Ocean View Internal Medicine, Long Beach, California
  - St Mary's Med Ctr, Long Beach, California
  - AIDS Healthcare Foundation-Research Center, Los Angeles, California
  - Kaiser Permanente LAMC, Los Angeles, California
  - LAC / USC Med Ctr / Infectious Diseases, Los Angeles, California
  - Cedars Sinai Med Ctr, Los Angeles, California
  - Tower Infectious Diseases / Med Associates Inc, Los Angeles, California
  - Robert Scott MD, Oakland, California
  - UCSD Med Ctr - Owen Clinic, San Diego, California
  - Pacific Horizons Med Group, San Francisco, California
  - Kaiser Foundation Hospital, San Francisco, California
  - San Francisco VA Med Ctr, San Francisco, California
  - Harbor UCLA Med Ctr / Research and Educational Institute, Torrance, California
  - Univ of Colorado / Health Science Ctr, Denver, Colorado
  - Yale New Haven Hosp / Nathan Smith Clinic, New Haven, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Physicans Home Service, Washington D.C., District of Columbia
  - Therafirst Med Ctr, Fort Lauderdale, Florida
  - ARTCTC, Ft. Pierce, Florida
  - Steinhart Medical Associates, Miami, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Hillsborough County Health Dept, Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - AIDS Research Consortium of Atlanta Inc, Atlanta, Georgia
  - Ponce de Leon Med Ctr, Atlanta, Georgia
  - Northstar Med Clinic, Chicago, Illinois
  - Bendel Med Research, Lafayette, Louisiana
  - Dr Joel Gallant, Baltimore, Maryland
  - New England Med Ctr, Boston, Massachusetts
  - Massachusetts Gen Hosp, Boston, Massachusetts
  - Harper Hosp, Detroit, Michigan
  - Regions Hosp / HIV/AIDS Program, Saint Paul, Minnesota
  - Univ of NM, Albuquerque, New Mexico
  - Albany Med College, Albany, New York
  - Brookdale Univ Hosp and Med Ctr, Brooklyn, New York
  - Howard Grossman, New York, New York
  - St Vincent's Hosp, New York, New York
  - Columbia Univ, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Nalle Clinic / Clinical Research Dept, Charlotte, North Carolina
  - Ian Baird, Columbus, Ohio
  - Remington Davis Inc, Columbus, Ohio
  - Oklahoma Univ Health Science Ctr, Oklahoma City, Oklahoma
  - Pennsylvania State College of Medicine, Hershey, Pennsylvania
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Dallas Veterans Administration Med Ctr, Dallas, Texas
  - Nicholas Bellos, Dallas, Texas
  - Thomas Street Clinic, Houston, Texas
  - Univ of Texas / Thomas Street Clinic, Houston, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Infectious Diseases Physicians Inc, Annandale, Virginia
  - Hampton Roads Med Specialists, Hampton, Virginia
  - Infections Ltd PS, Puyallup, Washington
  - Infections Ltd / Physicians Med Ctr, Tacoma, Washington
- Puerto Rico (3):
  - Ponce Univ Hosp, Ponce
  - Clinical Research Puerto Rico Inc, San Juan
  - San Juan AIDS Program, Santurce